CLINICAL TRIAL: NCT04656574
Title: The Effects of Mıxed Sımulatıon Traınıng Used in Vagınal Chıldbırth Wıth Epısıotomy on Student Medıcal Malpractıce Tendency And Perceptıons of Care Behavıors
Brief Title: The Effects of Sımulatıon Used in Vagınal Chıldbırth on Malpractıce Tendency And Perceptıons of Care Behavıors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Durmaz (Other)
Responsible Party: Sponsor-Investigator, Aysegul Durmaz, Asst. Prof., Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Sim. Malp. Percep.
Record Dates: First submitted 2020-11-28; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Behavior; Perceptions
Keywords: Episiotomy; Medical Malpractice; Perceptions; Simulation; Vaginal Childbirth
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: The study was conducted as a single blind, prospective, and simple randomized controlled trial. A power calculation was performed and with a standard deviation of 0.25 and statistical significance of 0.05, the number of students needed to total participate was determined to be 116, 58 per group. Out of 79 students, 60 were randomly assigned to the experimental group receiving education using simulation-based training and out of 90 students, 60 were randomly assigned to the control group that received the course explaining vaginal delivery for the first time.
Who Masked: Participant
Masking Description: Participants didn't know which group they were allocated. The participants will be blind when they receive simulation based training from researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental group received the course explaining vaginal delivery for the first timethat used simulation-based training.
  Interventions: Behavioral: Simulation-based training
- Control Group (No Intervention): Control group received the course explaining vaginal delivery for the first time

INTERVENTIONS:
Behavioral: Simulation-based training — The simulation training included the activities that midwives should do during the birth and management of vaginal delivery with episiotomy. The students received theoretical training, and to reinforce it, they were asked to mold a fetal head from a potato, make a cardboard cervix showing dilatation measurements during vaginal delivery, and make a fetal position identification model taking the occiput as a reference point.
  Arms: Experimental Group

SUMMARY:
H1a: The simulation-based training used to provide delivery skills have an effect on malpractice trends of midwifery students.

H1b: The simulation-based training used to provide delivery skills have an effect on midwifery students' perceptions of care behaviors.

H0a: The simulation-based training used to provide delivery skills have not an effect on malpractice trends of midwifery students.

H0b: The simulation-based training used to provide delivery skills have not an effect on midwifery students' perceptions of care behaviors.

DETAILED DESCRIPTION:
The study was conducted as a single blind, prospective, and simple randomized controlled trial. The study was conducted in the fall semester of 2016 and in the fall semester of 2017 in the midwifery department of a university.

The study universe comprised 79 students who took the course about vaginal delivery (which is included in the midwifery curriculum) provided using simulation-based training and 90 students taking this course for the first time. The study included 120 participants, including 60 randomly selected students who agreed to participate in the study, were enrolled in midwifery, and took the course explaining vaginal delivery for the first time and 60 randomly selected students who received this education using simulation-based training.

The simulation training included the activities that midwives should do during the birth and management of vaginal delivery. Bone pelvis, fetal head, fetus, cervical dilatation-effacement, fetal descensus, maternal-neonatal birthing simulators and chicken breast model for episiotomy were used by the researchers to monitor, manage, and provide care for the progress of labor. The students in the control group received theoretical training about management and care of vaginal delivery. In addition, the researchers demonstrated them how to monitor and manage the delivery process and provide care.

Data collection tools included a personal information form, medical malpractice tendency scale in nursing, and caring assessment questionnaire.

Statistical analyses were made using Statistical Package for Social Sciences (IBM SPSS) Statistics 22 software. The findings were analyzed using descriptive statistics (average, standard deviation, frequency, and percentage). The Kolmogorov-Smirnov test was used to determine normal distribution of the data.

ELIGIBILITY:
Inclusion Criteria:

* To receive simulation based training
* Older than 18 years,
* To Voluntary to participate,
* To know how to read, write and speak in Turkish,
* To do model work
* Fully completed the data collection forms
* To continue the all course

Exclusion Criteria:

* To received theoretical training,
* Younger than 18 years,
* Refuse to participate
* Not knowing how to read, write and speak Turkish,
* Not to do model work
* Not to fill the questionnaire
* Not to continue the course

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-01-07 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
medical malpractice tendency | 2 week after the intervention
  The medical malpractice tendency scale in nursing includes routine patient care activities of the nurses. It was developed by Özata and Altunkan (14). The Likert-type scale, scored between 1 and 5, includes 49 items and consists of five subscales. The scoring is 1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always. The minimum score is 49 and maximum is 245 points. A higher total score indicates that nurses have less medical malpractice tendencies. The scale includes five subscales: drug and transfusion administration, prevention of infections, patient monitıring and material-device safety, prevention of falls, and communication.
Perceptions of care behaviors | 2 week after the intervention
  Caring Assessment Questionnaire/Care-Q scale: The caring assessment questionnaire/Care-Q was developed by Lee, Larson, and Holzemer (18) and adapted to Turkish by Eskimez and Acaroğlu (19). This Likert-type scale, scored between 1 and 7, includes 50 items and consists of six subscales. The scoring is 1=Never, 2=Rarely, 3=Occasionally, 4=Sometimes, 5=Frequently, 6=Usually, 7=Every time. The minimum score is 50 and maximum is 350 points. A higher score indicates a positive increase in the frequency of providing and perceiving care behaviors. The six subscales are attainability, descriptions and facilities, comfort, expectations, reassuring communication, and observation and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Durmaz, Principal Investigator — KSBU
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: If study IPD is used, my article should be cited.

REFERENCES:
- [Result] Dearnley CA, Meddings FS. Student self-assessment and its impact on learning - a pilot study. Nurse Educ Today. 2007 May;27(4):333-40. doi: 10.1016/j.nedt.2006.05.014. Epub 2006 Jul 25. PMID 16870309
- [Result] Valen K, Holm AL, Jensen KT, Grov EK. Nursing students' perception on transferring experiences in palliative care simulation to practice. Nurse Educ Today. 2019 Jun;77:53-58. doi: 10.1016/j.nedt.2019.03.007. Epub 2019 Mar 30. PMID 30954856
- [Result] Lendahls L, Oscarsson MG. Midwifery students' experiences of simulation- and skills training. Nurse Educ Today. 2017 Mar;50:12-16. doi: 10.1016/j.nedt.2016.12.005. Epub 2016 Dec 16. PMID 28006699
- [Result] Doody O, Condon M. Using a simulated environment to support students learning clinical skills. Nurse Educ Pract. 2013 Nov;13(6):561-6. doi: 10.1016/j.nepr.2013.03.011. Epub 2013 Apr 18. PMID 23602694
- [Result] Posmontier B, Montgomery K, Smith Glasgow ME, Montgomery OC, Morse K. Transdisciplinary teamwork simulation in obstetrics-gynecology health care education. J Nurs Educ. 2012 Mar;51(3):176-9. doi: 10.3928/01484834-20120127-02. Epub 2012 Jan 27. PMID 22283152
- [Result] Miles DA. Simulation Learning and Transfer in Undergraduate Nursing Education: A Grounded Theory Study. J Nurs Educ. 2018 Jun 1;57(6):347-353. doi: 10.3928/01484834-20180522-05. PMID 29863735
- [Result] Cantrell ML, Meyer SL, Mosack V. Effects of Simulation on Nursing Student Stress: An Integrative Review. J Nurs Educ. 2017 Mar 1;56(3):139-144. doi: 10.3928/01484834-20170222-04. PMID 28263351
- [Result] Landeen J, Pierazzo J, Akhtar-Danesh N, Baxter P, van Eijk S, Evers C. Exploring Student and Faculty Perceptions of Clinical Simulation: A Q-Sort Study. J Nurs Educ. 2015 Sep;54(9):485-91. doi: 10.3928/01484834-20150814-02. PMID 26334334
- [Result] Guler H, Cetin P, Yurtsal ZB, Cesur B, Bekar M, Ucar T, Evcili F, Cetin A. Effect of episiotomy training with beef tongue and sponge simulators on the self-confidence building of midwifery students. Nurse Educ Pract. 2018 May;30:1-6. doi: 10.1016/j.nepr.2018.02.004. Epub 2018 Feb 9. PMID 29452943